CLINICAL TRIAL: NCT01316679
Title: An Analysis of Urinary Proteases as Biomarkers for Hepatocellular Carcinoma-101423
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David L Gorden, Professor, Vanderbilt University Medical Center
Other Study IDs: Urinary Biomarkers 101423
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma; Liver Disease
Keywords: HCC; Liver Disease without HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group A: Patients with known HCC
- Group B: Patients with liver disease but no HCC
- Group C: Control; patients with no known liver disease or HCC

SUMMARY:
Specific urine proteases or groups of these enzymes can be reliable biomarkers and an effective gauge of response to therapy in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* Must be between 18-90 years of age at the time of consent
* Ability to provide urine specimen at protocol-defined timepoints
* Must have treatment interventions planned that are directly related to liver disease (excluding those assigned to group 3-Controls)

Exclusion Criteria:

* Suspected inability, e.g. unwillingness to comply with study procedures or unwillingness to provide written consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Vanderbilt internal medicine, hepatology, hepatobiliary surgery, and general surgery clinics.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)